CLINICAL TRIAL: NCT03579771
Title: A Single-Arm Feasibility Study of Gemcitabine, Cisplatin, and Nab-Paclitaxel as Neoadjuvant Therapy for Resectable Oncologically High-Risk Intrahepatic Cholangiocarcinoma
Brief Title: Gemcitabine, Cisplatin, and Nab-Paclitaxel Before Surgery in Patients With High-Risk Liver Bile Duct Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Celgene (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shishir Kumar Maithel, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00104175; NCI-2018-00998 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EU4339-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Resectable Cholangiocarcinoma; Stage IB Intrahepatic Cholangiocarcinoma AJCC v8; Stage II Intrahepatic Cholangiocarcinoma AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIA Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIB Intrahepatic Cholangiocarcinoma AJCC v8
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cisplatin; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine, cisplatin, nab-paclitaxel (Experimental): Participants receive nab-paclitaxel IV over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Participants with stable disease (SD), partial response (PR), or complete response (CR) then undergo standard of care hepatectomy with portal lymphadenectomy.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: CDDP; Cis-diamminedichloridoplatinum; Cismaplat; Cisplatinum; Neoplatin; Platamin; Platinol
Drug: Gemcitabine — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine hydrochloride; Gemcitabine hydrochloride; Gemzar
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI-007; Abraxane; Nanoparticle albumin-bound paclitaxel

SUMMARY:
This phase II trial studies how well gemcitabine, cisplatin, and nab-paclitaxel work before surgery in treating participants with high-risk bile duct cancer in the liver (intrahepatic cholangiocarcinoma). Drugs used in chemotherapy, such as nab-paclitaxel, cisplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To assess the feasibility of therapeutic approach that includes neoadjuvant chemotherapy including gemcitabine hydrochloride (gemcitabine), cisplatin, and nab-paclitaxel for high-risk but technically resectable intrahepatic cholangiocarcinoma and is completed with surgical resection.

SECONDARY OBJECTIVES:

I. To assess the radiological response rate to neoadjuvant systemic chemotherapy according to the Response Evaluation Criteria in Solid Tumors (RECIST).

II. To determine the R0 resection rate.

III. To determine patient recurrence-free survival (RFS).

IV. To identify patient overall survival (OS) rate.

OUTLINE:

Participants receive nab-paclitaxel intravenously (IV) over 30 minutes, cisplatin IV over 60 minutes, and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Participants with stable disease (SD), partial response (PR), or complete response (CR) then undergo standard of care hepatectomy with portal lymphadenectomy.

After completion of study treatment, participants are followed up every 4 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intrahepatic cholangiocarcinoma.
* High-quality cross-sectional imaging by computerized tomography (CT) or magnetic resonant imaging (MRI) performed within 6 weeks prior to enrollment and showed a resectable, but high-risk, intrahepatic cholangiocarcinoma (IHCCA) confined to the liver, bile duct, and/or regional lymph nodes. Tumors will be considered high-risk if the high-quality, contrast-enhanced CT and/or MRI +/- positron emission tomography (PET) scan showed: (must meet at least one of the criteria below)

  1. T-stage ≥ Ib (Ib-IV)
  2. Solitary lesion > 5 cm
  3. Multifocal tumors or satellite lesions present confined to the same lobe of the liver as the dominant lesion but still technically resectable
  4. Presence of major vascular invasion but still technically resectable
  5. Suspicious or involved regional lymph nodes (N1)
* No distant extrahepatic disease (M0)
* Able to give informed consent.
* Able to adhere to study visit schedule and other protocol requirements.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Absolute neutrophil count (ANC) ≥ 1,500 cells/μL
* Platelet count ≥ 100,000 cells/μL
* Hemoglobin ≥ 9 g/dL
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Albumin ≥ 3 g/dL
* Creatinine ≤ 1.5 x ULN
* Non-pregnant and non-lactating.
* Women of child-bearing potential (defined as a sexually mature woman who [1] has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must commit to true abstinence from heterosexual contact or agree to use, and be able to comply with, effective contraception without interruption for 28 days prior to starting gemcitabine/cisplatin/nab-paclitaxel (including dose interruptions) until treatment with gemcitabine/cisplatin/nab-paclitaxel is complete.
* Male subjects must practice true abstinence or agree to use a condom during sexual contact with a female of childbearing potential or a pregnant female while on treatment (including during dose interruptions) with gemcitabine/cisplatin/nab-paclitaxel and for 6 months following gemcitabine/cisplatin/nab-paclitaxel discontinuation, even if he has undergone a successful vasectomy.

Exclusion Criteria:

* Peripheral neuropathy of grade 2 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 4.0. In CTCAE version 4.0 grade 2 sensory neuropathy is defined as "moderate symptoms; limiting instrumental activities of daily living (ADLs)".
* Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, symptomatic congestive heart failure, uncontrolled diabetes, serious active, uncontrolled infection after inadequate biliary drainage if tumor obstructing bile duct, or psychiatric illness/social situations.
* Pregnancy (positive pregnancy test) or lactation.
* Known central nervous system (CNS) disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded.
* Previous (within the past 5 years) or concurrent presence of other cancer, except non-melanoma skin cancer and in situ carcinomas.
* History of allergy or hypersensitivity to any of the study drugs.
* Current abuse of alcohol or illicit drugs.
* Inability or unwillingness to sign the informed consent form.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shishir Maithel, MD, Principal Investigator — Emory University
Locations (7):
- United States (7):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
Started | 30
Completed | 22
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.17 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Benaroya Research Institute at Virginia Mason | 3
  Emory University | 11
  MD Anderson | 12
  Mayo Clinic-Rochester | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed All Preoperative and Operative Therapy
Description: Completion of all therapy rate will be recorded.
Time Frame: Up to 12 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
Number analyzed (Participants) | 30
Participants | 22

2. Primary Outcome: Number of Participants With Adverse Events
Description: Will be monitored using method of Thall, Simon and Estey, and will be tabulated by the maximum reported Common Terminology Criteria for Adverse Events (CTCAE) grade.
Time Frame: Up to 3 years after study start
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
Number analyzed (Participants) | 30
participants
  Any adverse event | 26
  Blood and lymphatic system disorders | 13
  Ear and labyrinth disorders | 2
  Endocrine disorders | 1
  Gastrointestinal disorders | 11
  General disorders and administration site conditions | 11
  Investigations | 15
  Metabolism and nutrition disorders | 4
  Nervous system disorders | 9
  Renal and urinary disorders | 1
  Respiratory, thoracic and mediastinal disorders | 4
  Skin and subcutaneous tissue disorders | 13
  Vascular disorders | 1

3. Secondary Outcome: Radiological Response Rate Defined as the Percentage of Patients Who Will Have Complete Response (CR), Partial Response (PR) or Stable Disease (SD) After the Neoadjuvant Therapy
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 12 weeks after study start
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
Number analyzed (Participants) | 30
Participants
  PD | 3
  PR | 7
  SD | 20

4. Secondary Outcome: Recurrence-free Survival (RFS)
Description: RFS is defined as the time between the date of surgery and the date of disease recurrence or death, whichever occurred first. If a patient did not have an event (i.e. disease recurrence or death) by the time of final analysis, patient will be censored at the last disease evaluation time.
Time Frame: From the date of surgery up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
Number analyzed (Participants) | 30
months | 23.7 [17.1 to 37.1]

5. Secondary Outcome: Number of Participants With Overall Survival
Description: OS is defined as the time from date of neoadjuvant treatment start to the date of death from any cause or to the date of last follow-up if patients are alive. If a patient is alive by the time of final analysis, the patient will be censored at the last follow-up date.
Time Frame: From date of neoadjuvant treatment start up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Gemcitabine, Cisplatin, Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine, Cisplatin, Nab-paclitaxel (N=30)
Anemia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Neutrophil count decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dehydration (General disorders) | 1
Hypophosphatemia (Investigations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine, Cisplatin, Nab-paclitaxel (N=30)
Fatigue (General disorders) | 20
Abdominal pain (Gastrointestinal disorders) | 13
Anemia (Blood and lymphatic system disorders) | 13
Diarrhea (Gastrointestinal disorders) | 13
Hyperglycemia (Endocrine disorders) | 12
Neutrophil count decreased (Blood and lymphatic system disorders) | 12
Nausea (Gastrointestinal disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 10
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 9
Constipation (Gastrointestinal disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 8
Platelet count decreased (Blood and lymphatic system disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
White blood cell decreased (Blood and lymphatic system disorders) | 8
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 7
Anorexia (Gastrointestinal disorders) | 6
General disorders and administration site conditions - Other, specify (General disorders) | 6
Hyponatremia (Blood and lymphatic system disorders) | 6
Anxiety (Psychiatric disorders) | 5
Aspartate aminotransferase increased (Investigations) | 5
Dizziness (General disorders) | 5
Dyspnea (Gastrointestinal disorders) | 5
Hypertension (Cardiac disorders) | 5
Insomnia (Psychiatric disorders) | 5
Pain (General disorders) | 5
Blurred vision (Eye disorders) | 4
Edema limbs (Blood and lymphatic system disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hypokalemia (Investigations) | 3
Hypomagnesemia (Blood and lymphatic system disorders) | 3
Mucositis oral (Infections and infestations) | 3
Tinnitus (Ear and labyrinth disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Creatinine increased (Investigations) | 2
Epistaxis (Ear and labyrinth disorders) | 2
Febrile neutropenia (Infections and infestations) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hypotension (Cardiac disorders) | 2
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Sore throat (Infections and infestations) | 2
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Bronchial infection (Ear and labyrinth disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chills (General disorders) | 1
Colitis (Infections and infestations) | 1
Cough (Infections and infestations) | 1
Dehydration (General disorders) | 1
Depression (Psychiatric disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Erythema multiforme (Blood and lymphatic system disorders) | 1
Flushing (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (General disorders) | 1
Hypercalcemia (Blood and lymphatic system disorders) | 1
Hyperkalemia (Blood and lymphatic system disorders) | 1
Hypoglycemia (Endocrine disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Injection site reaction (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Investigations - Other, specify (Investigations) | 1
Laryngeal inflammation (Ear and labyrinth disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Localized edema (Injury, poisoning and procedural complications) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Movements involuntary (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Myalgia (General disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Pulmonary hypertension (Cardiac disorders) | 1
Renal and urinary disorders - Other, specify (Endocrine disorders) | 1
Renal colic (Endocrine disorders) | 1
Sick sinus syndrome (Ear and labyrinth disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urine discoloration (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03579771/Prot_SAP_002.pdf
  • Informed Consent Form (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03579771/ICF_000.pdf